CLINICAL TRIAL: NCT02874924
Title: Effect of Mammalian Target of Rapamycin Inhibition and Other Metabolism Modulating Interventions on the Elderly: Immune, Cognitive, and Functional Consequences
Brief Title: Effect of mTOR Inhibition and Other Metabolism Modulating Interventions on the Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HSC20120304H
Record Dates: First submitted 2016-06-14; First posted 2016-08-22 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-03

CONDITIONS: Aging
Keywords: Geriatrics
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rapamycin (Experimental): Rapamycin 1mg taken once daily for 8 weeks
  Interventions: Drug: Rapamycin
- Placebo (Placebo Comparator): Placebo taken once daily for 8 weeks
  Interventions: Drug: Placebo
- Rapamycin Alone - Cardiovascular Effects (Experimental): No placebo control; Rapamycin 1mg once daily for 8 weeks
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — treatment
  Other Names: Sirolimus
  Arms: Rapamycin
Drug: Placebo — control
  Arms: Placebo
Drug: Rapamycin — No placebo control in this substudy group
  Other Names: Sirolimus
  Arms: Rapamycin Alone - Cardiovascular Effects

SUMMARY:
The ability to mount an effective immune response declines with age, leaving the elderly increasingly susceptible to infectious diseases and cancer. Rapamycin, an FDA approved drug to prevent transplant rejection, increases the lifespan and healthspan of mice and ameliorates age-related declines in immune responsiveness, cancer survival, and cognition in laboratory animals. Investigators are conducting a translational trial to test whether rapamycin also improves life functions in humans focusing on elderly persons (aged 70-95).

DETAILED DESCRIPTION:
Inhibition of the mTOR pathway by rapamycin (RAPA), an immunosuppressive drug used as adjunct therapy in preventing solid organ allograft rejection, enhances longevity in mice. Importantly, RAPA was efficacious even when initiated in relatively old animals. Thus, it has been suggested that RAPA could be used therapeutically in humans to slow age-associated pathologies. Indeed, improvements in cognition, control of tumorigenesis, and enhancing certain aspects of immunity have been demonstrated in RAPA treated murine models. Moreover, long-term RAPA delivery in older mice is associated with changes in immune reactivity not evident in younger animals. Investigators propose to expand to a larger cohort of older humans to test the hypothesis that RAPA treatment, even in very old individuals, will result in simultaneous improvement in systems known to be negatively affected by aging. Investigators will focus on the immune system, cognition, and physical parameters of healthy aging, such as walking speed. Investigators will recruit healthy volunteers, aged 75-95 years, and randomize them to either RAPA or placebo, controlling for gender, ethnicity, and age. These groups will be used to address the following specific aims: Aim 1. Assess general parameters of immune health before and after RAPA treatment; these include serum inflammatory cytokines, PBMC subsets (naïve vs memory T cells, TREGS, etc.), and polyclonal T cell activation potential. Aim 2. Test the effects of RAPA treatment on responsiveness to a vaccine challenge; both B cell (antibody) and T cell responses will be assessed. Aim 3. Correlate immune function rejuvenation with cognitive and physical function measures in subjects treated with RAPA or placebo. Aim 4. Collect pilot data on effect of RAPA on cardiovascular function. Cognition will be assessed by three different testing tools (EXIT25, SLUMS, and TAPS). Physical performance will be measured by grip strength and 40 foot timed walks, parameters known to correlate with healthy aging. Measures of cardiovascular function (Substudy D) using MRI of the heart to evaluate diastolic function and brain MRI to analyze cerebral blood flow, with measures of pulse wave velocity and endothelial function using laser doppler flowmetry will be performed. In addition to scoring positive outcomes, investigators will assess whether there are adverse changes in clinical laboratory tests that could compromise the safe use of RAPA therapeutically in older individuals. The long-term goal is to assess whether RAPA is safe to use in an elderly population, while also being efficacious in slowing, or even reversing, the aging process.

ELIGIBILITY:
Inclusion Criteria: age 70-95

* participants will be in good health with all chronic diseases (hypertension, coronary artery disease, etc.) clinically stable.
* participants must have adequate cognitive function to be able to give informed consent. This will be established by enrolling participants with CLOX 1 scores of ≥10.

Exclusion Criteria:

* unstable ischemic heart disease
* clinically significant pulmonary disease
* history of immunodeficiency or receiving immunosuppressive therapy
* history of a coagulopathy or receiving a medical condition requiring anticoagulation
* an estimated glomerular filtration rate of <30ml/min
* uncontrolled hypercholesteremia >350mg/dl;
* uncontrolled hypertriglyceridemia >500mg/dl
* diabetes
* history of skin ulcers or poor wound healing
* smoking
* liver disease
* treatment with drugs known to affect cytochrome P450 3A (diltiazem, erythromycin)

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Kellogg, MD PhD, Principal Investigator — University of Texas
Locations (1):
- UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
Started | 14 | 14 | 6
Completed | 11 | 14 | 6
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects | Total
Number analyzed (Participants) | 14 | 14 | 6 | 34
Age, Customized [Count of Participants; unit: Participants] — Only participants age 70 years or older were eligible
  Participants
    Age, 70 years and older | 14 | 14 | 6 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 0 | 10
  Male | 9 | 9 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 1 | 10
  Not Hispanic or Latino | 7 | 12 | 5 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 14 | 6 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 6 | 34

OUTCOME MEASURES:

1. Primary Outcome: Immunological Responses
Description: T cell function measured by number of T cells per millimeter cubed.
Time Frame: 8 weeks
Population: In the cardiovascular arm, no T cell function was analyzed.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
Number analyzed (Participants) | 11 | 14 | 0
cells/mm^3 | 8.33 (3.82) | 11.24 (4.45) |
Statistical Analysis 1: Comparison: Rapamycin vs Placebo; Null hypothesis; Test type: Equivalence — Pilot study, therefore, no power calculation available; p = 0.56, t-test, 2 sided; Mean Difference (Net) = -1.81, 95% CI 2-sided [-8.48 to 4.86]

2. Secondary Outcome: Physical Performance
Description: walking speed: Timed 40-foot walk: each participant will perform 3 walks (timed with a stopwatch) at their preferred walking speed over a measured 40-foot path. Results will be averaged for analysis. The faster the walking speed the better the performance.
Time Frame: 8 weeks
Population: Walking speed was not analyzed in the cardiovascular group.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
Number analyzed (Participants) | 11 | 14 | 0
Seconds | 7.75 (1.12) | 7.17 (1.12) |

3. Secondary Outcome: Cognitive Function
Description: The Executive Interview (EXIT25) - This test is a brief bedside test that consists of 25 items measuring abilities that include:
  Executive functioning, Motor sequencing, Spoken alternate sequencing, Verbal fluency, Design fluency, Persistence, Resistance to interference, Reflexes Scoring directions are listed under each of the 25 portions of this test. For each section, the client is given a score of a 0, 1, or 2. A score "0" indicates no impairment, a score of "1" indicates some impairment, and a score of "2" indicates severe impairment. Directions for what qualifies as each score are listed under each section. The points are totaled and criteria are given for severe, moderate, and no impairment. Minimum score is -0- and maximum is 50. A score of 15 or below indicates normal executive functioning, a score of above 15 indicates moderate to severe impairment.
Time Frame: 8 weeks
Population: EXIT25 was not collected or analyzed in cardiovascular group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
Number analyzed (Participants) | 14 | 14 | 0
score on a scale | 7.2 (4.52) | 6.92 (4.23) |

4. Other Pre Specified Outcome: Cardiovascular Effect
Description: Pulse Wave Velocity is measured using an Electrocardiogram (ECG)
Time Frame: 8 weeks
Population: Due to technical problems with equipment, data were not captured for analysis.
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
Number analyzed (Participants) | 0 | 0 | 0

5. Other Pre Specified Outcome: Volume of Diastolic Filling
Description: Diastolic function was assessed using Magnetic Resonance Imaging (MRI) of the heart to measure the diastolic filling of the heart in participants in the open label rapamycin group.
Time Frame: 8 weeks
Population: Cardiovascular effects were not measured in the Rapamycin versus placebo group, only open label rapamycin group.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
Number analyzed (Participants) | 0 | 0 | 6
milliliters |  |  | 132.84 (26.82)

ADVERSE EVENTS:
Time Frame: 8 weeks per subject
Arm/Group | Rapamycin | Placebo | Rapamycin Alone - Cardiovascular Effects
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 2/14 | 0/14 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rapamycin (N=14) | Placebo (N=14) | Rapamycin Alone - Cardiovascular Effects (N=6)
Rash of face (General disorders) | 1 (1) | 0 (0) | 0 (0) — Acneform rash
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT02874924/Prot_SAP_000.pdf